CLINICAL TRIAL: NCT02287402
Title: Postmarketing Clinical Study on AO-128
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AO-128/OCT-910; JapicCTI-101004 (Other: JapicCTI); U1111-1163-1618 (Registry Identifier: WHO)
Record Dates: First submitted 2014-10-22; First posted 2014-11-10 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Impaired Glucose Tolerance (IGT)
MeSH Terms: conditions — Glucose Intolerance | interventions — AO 128; voglibose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AO-128 0.6 mg (Experimental): One AO-128 0.2 mg tablet was taken orally 3 times a day before meals.
  Interventions: Drug: AO-128

INTERVENTIONS:
Drug: AO-128 — AO-128 tablet
  Other Names: Voglibose; BASEN

SUMMARY:
The purpose of open-label study is to evaluate the efficacy and safety of AO-128 (Voglibose) 0.6 mg/day in patients with impaired glucose tolerance (IGT) who had been non-responsive to diet therapy and exercise therapy, and follow up the progress after the end of treatment in patients who was assessed as normoglycemic.

DETAILED DESCRIPTION:
The α-glucosidase inhibitor voglibose was developed by Takeda Pharmaceutical Co. Ltd and is one of the most commonly used oral antidiabetic agents in Japan. Voglibose is used as first-line treatment for improvement of postprandial hyperglycemia in diabetic patients with inadequate response to diet and exercise therapy and as add-on treatment to other oral antidiabetic drugs and insulin. In 2009, voglibose was approved in Japan for the management of prediabetes (IGT).

This study was a single-group, multi-center, open-label study. The study period consisted of a screening period of 1 week or less, a treatment period of 96 weeks or more, and a follow-up period of 48 weeks. However, if a patient was assessed as having type 2 diabetes mellitus or normoglycemia, the treatment period was to be ended, and only those assessed as normoglycemic were to proceed to follow-up. Follow-up was also to be terminated if patients were assessed as having IGT or type 2 diabetes mellitus during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on diet therapy and exercise therapy for 3 to 6 months prior to the start of screening, with baseline (fasting ) plasma glucose < 126 mg/dL and 2-hour plasma glucose of 140 to 199 mg/dL (revised WHO criteria) during a 75 g oral glucose tolerance test (OGTT) in the screening period
2. Patients meeting any of 1 through 4 below:

   * 1) Comorbid hypertension or high normal blood pressure
   * 2) Comorbid dyslipidemia
   * 3) Comorbid obesity
   * 4) Patients with up to a second-degree family history of type 2 diabetes mellitus
3. Patients with HbA1c < 6.5% in the screening period
4. Male or female patients at least 20 years of age at the time informed consent was obtained
5. Treatment category: Outpatient

Exclusion Criteria:

1. Patients previously diagnosed with diabetes mellitus.
2. Patients with apparent impaired glucose metabolism or with a disease or condition potentially involving impaired glucose metabolism.
3. Patients with serious hepatic impairment.
4. Patients with serious renal impairment.
5. Patients with serious cardiac, cerebrovascular, pancreatic, hematologic, or other disease.
6. Patients with a history of intestinal obstruction or a history of laparotomy within 6 months (24 weeks) before the start of screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 30 investigative sites in Japan from 9 March 2010 to 15 November 2012.
Pre-assignment Details: Participants with impaired glucose tolerance (IGT) who had been non-responsive to diet therapy and exercise therapy receive one AO-128 0.2 mg tablet orally 3 times a day before meals.
Period: Treatment Period
Arm/Group | AO-128 0.6 mg
Started | 197
Completed | 170
Not Completed | 27
Not completed — Adverse Event | 17
Not completed — Voluntary Withdrawal | 10
Period: Follow-up
Arm/Group | AO-128 0.6 mg
Started | 106 (64 participants who completed the Treatment Period did not continue to Follow-up.)
Completed | 103
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Voluntary Withdrawal | 2

BASELINE CHARACTERISTICS:
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.35)
Age, Customized [Number; unit: participants]
  <65 years | 137
  ≥65 years | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 129
Region of Enrollment [Number; unit: participants]
  Japan | 197

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Diabetic Status in the Treatment Period (Type 2 Diabetes Mellitus, Normoglycemia, or Impaired Glucose Tolerance (IGT)
Description: Frequency tabulations of the "assessment of diabetic status in the treatment period (Type 2 Diabetes mellitus, normoglycemia, or IGT)" were prepared in the "Full Analysis Set".
Time Frame: Treatment period: Up to 122 weeks. Treatment was to be ended when patients were assessed as Type 2 Diabetes Mellitus or normoglycemic.
Population: Full Analysis Set - All participants who received at least 1 dose of open-label study drug.
Measure: Number; unit: participants
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 197
participants
  Type 2 Diabetes mellitus | 25
  Normoglycemia | 106
  IGT | 66

2. Primary Outcome: Assessment of Diabetic Status in Follow-up (Type 2 Diabetes Mellitus, Normoglycemia, or IGT)
Description: Frequency tabulations of the "assessment of diabetic status in the follow-up (Type 2 Diabetes mellitus, normoglycemia, or IGT)" were prepared in patients who proceeded to the follow-up in the "Full Analysis Set".
Time Frame: Follow-up at Week 12, 24, 36, and 48
Population: Participants from the Full Analysis Set, all participants who received at least 1 dose of open-label study drug, and continued to Follow-up.
Measure: Number; unit: participants
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 106
participants
  Type 2 Diabetes mellitus | 3
  Normoglycemia | 9
  IGT | 94

3. Secondary Outcome: Time to Progression to Type 2 Diabetes Mellitus in the Treatment Period Calculated by the Kaplan-Meier Method
Description: The cumulative progression rate (percentage of participants) was calculated by the Kaplan-Meier method for the "time to progression to Type 2 Diabetes mellitus in the treatment period" in the "Full Analysis Set".
Time Frame: Day 168, 336, 504, and 672
Population: Full Analysis Set - All participants who received at least 1 dose of open-label study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 197
percentage of participants
  Day 168 | 0.0
  Day 336 | 4.4
  Day 504 | 10.2
  Day 672 | 16.9

4. Secondary Outcome: Time to Progression to Type 2 Diabetes Mellitus in the Treatment Period Calculated Using the Cumulative Incidence Function
Description: The cumulative progression rate (percentage of participants) was calculated using the cumulative incidence function for the "time to progression to type 2 diabetes mellitus in the treatment period" in the "Full Analysis Set".
Time Frame: Day 168, 336, 504, and 672
Population: Full Analysis Set - All participants who received at least 1 dose of open-label study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 197
percentage of participants
  Day 168 | 0.0
  Day 336 | 3.3
  Day 504 | 6.9
  Day 672 | 10.0

5. Secondary Outcome: Time to Improvement to Normoglycemia in the Treatment Period Calculated by the Kaplan-Meier Method
Description: The cumulative progression rate (percentage of participants) was calculated by the Kaplan-Meier method for the "time to improvement to normoglycemia in the treatment period" in the "Full Analysis Set".
Time Frame: Day 168, 336, 504, and 672
Population: Full Analysis Set - All participants who received at least 1 dose of open-label study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 197
percentage of participants
  Day 168 | 18.9
  Day 336 | 37.5
  Day 504 | 50.2
  Day 672 | 60.3

6. Secondary Outcome: Time to Improvement to Normoglycemia in the Treatment Period Measured Values by the Cumulative Incidence Function
Description: The cumulative progression rate (percentage of participants) was calculated using the cumulative incidence function for the "time to improvement to normoglycemia in the treatment period" in the "Full Analysis Set".
Time Frame: Day 168, 336, 504, and 672
Population: Full Analysis Set - All participants who received at least 1 dose of open-label study drug.
Measure: Number; unit: percentage of participants
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 197
percentage of participants
  Day 168 | 18.9
  Day 336 | 36.9
  Day 504 | 48.4
  Day 672 | 57.1

7. Secondary Outcome: 2-Hour Plasma Glucose During 75 g Oral Glucose Tolerance Test (OGTT)
Description: Summary statistics were calculated at each assessment time point for the 2-hour plasma glucose during 75 g OGTT in the "Full Analysis Set."
Time Frame: Week 0, 24, 48, 72, 96, 120, and the end of the treatment period
Population: Full Analysis Set - All participants who received at least 1 dose of open-label study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 197
mg/dL
  Week 0 | 166.7 (17.34)
  Week 24 | 148.0 (34.30)
  Week 48 | 153.2 (36.58)
  Week 72 | 155.6 (36.77)
  Week 96 | 155.6 (33.17)
  Week 120 | 163.2 (31.89)
  The end of the treatment period | 142.8 (37.73)

8. Secondary Outcome: 2-Hour Plasma Glucose During 75 g OGTT at Follow-up
Description: Summary statistics were calculated at each assessment time point for the 2-hour plasma glucose during 75 g OGTT in participants who proceeded to the follow-up in the "Full Analysis Set."
Time Frame: Follow-up at week 0, 12, 24, 36, and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 106
mg/dL
  Follow-up at Week 0 | 119.4 (15.82)
  Follow-up at Week 12 | 148.3 (35.26)
  Follow-up at Week 24 | 147.9 (29.69)
  Follow-up at Week 36 | 145.9 (18.94)
  Follow-up at Week 48 | 138.3 (20.06)

9. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: Summary statistics were calculated at each assessment time point for the HbA1c in the "Full Analysis Set."
Time Frame: Week 0, 12, 24, 48, 72, 96, 120, and the end of the treatment period.
Population: Full Analysis Set - All participants who received at least 1 dose of open-label study drug.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 197
percent
  Week 0 | 5.45 (0.331)
  Week 12 | 5.35 (0.305)
  Week 24 | 5.30 (0.302)
  Week 48 | 5.37 (0.317)
  Week 72 | 5.34 (0.285)
  Week 96 | 5.41 (0.269)
  Week 120 | 5.45 (0.256)
  The end of the treatment period | 5.35 (0.323)

10. Secondary Outcome: HbA1c at Follow-up
Description: Summary statistics were calculated at each assessment time point for the HbA1c in patients who proceeded to the follow-up in the "Full Analysis Set."
Time Frame: Follow-up at Week 0, 12, 24, 36, and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 106
percent
  Follow-up at Week 0 | 5.23 (0.292)
  Follow-up at Week 12 | 5.27 (0.330)
  Follow-up at Week 24 | 5.26 (0.326)
  Follow-up at Week 36 | 5.20 (0.301)
  Follow-up at Week 48 | 5.28 (0.260)

11. Secondary Outcome: Body Weight
Description: Summary statistics were calculated at each assessment time point for the body weight in the "Full Analysis Set."
Time Frame: Week 0, 12, 24, 48, 72, 96, 120, and the end of the treatment period
Population: Full Analysis Set - All participants who received at least 1 dose of open-label study drug.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 197
kg
  Week 0 | 70.74 (13.708)
  Week 12 | 69.74 (13.659)
  Week 24 | 69.91 (13.658)
  Week 48 | 69.25 (13.632)
  Week 72 | 70.03 (13.955)
  Week 96 | 69.25 (14.484)
  Week 120 | 68.82 (14.835)
  The end of the treatment period | 68.96 (13.892)

12. Secondary Outcome: Body Weight at Follow-up
Description: as for outcome 10
Time Frame: Follow-up at Week 0, 12, 24, 36, and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | AO-128 0.6 mg
Number analyzed (Participants) | 106
kg
  Follow-up at Week 0 | 67.60 (13.023)
  Follow-up at Week 12 | 67.76 (13.035)
  Follow-up at Week 24 | 68.87 (11.703)
  Follow-up at Week 36 | 70.13 (11.754)
  Follow-up at Week 48 | 68.72 (13.844)

ADVERSE EVENTS:
Time Frame: From the first dose of open-label study drug until the day of the last dose of open-label study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | AO-128 0.6 mg
Serious Adverse Events (participants affected / at risk) | 15/197
Other Adverse Events (participants affected / at risk) | 165/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AO-128 0.6 mg (N=197)
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Herpes zoster oticus (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nystagmus (Nervous system disorders) | 1
Cataract (Eye disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Calculus urinary (Renal and urinary disorders) | 2
Calculus ureteric (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AO-128 0.6 mg (N=197)
Nasopharyngitis (Infections and infestations) | 52
Influenza (Infections and infestations) | 8
Pharyngitis (Infections and infestations) | 7
Bronchitis (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 6
Seasonal allergy (Immune system disorders) | 7
Headache (Nervous system disorders) | 7
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 29
Flatulence (Gastrointestinal disorders) | 28
Abdominal distension (Gastrointestinal disorders) | 26
Constipation (Gastrointestinal disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Alanine aminotransferase increased (Investigations) | 6
Contusion (Injury, poisoning and procedural complications) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.